CLINICAL TRIAL: NCT01630226
Title: Cisplatin-monotherapy in the Treatment of BRCA1 Positive Breast Cancer Patients in Poland
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: Maria Sklodowska-Curie National Research Institute of Oncology (Other); Regional Oncology Hospital, Bielsko-Biala, Poland (Unknown)
Responsible Party: Principal Investigator, Tomasz Byrski, MD, PhD, MD, PhD, Pomeranian Medical University Szczecin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN-001/83/07-B
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: BRCA1 Mutation; Breast Cancer Invasive Nos
Keywords: BRCA1; pathological complete response; neoadjuvant chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant Cisplatin Chemotherapy (Experimental)
  Interventions: Drug: Neoadjuvant Cisplatin Chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant Cisplatin Chemotherapy — Patients will be treated with cisplatin chemotherapy at a dose of 75mg/m2 every three weeks for a total of four cycles (4 cycles of neoadjuvant chemotherapy).

SUMMARY:
This is a single center, non-randomized, open label phase II trial to evaluate the clinical and pathologic response of neoadjuvant cisplatin-monotherapy in BRCA1 positive patients. The study will enroll patients with diagnosed breast cancer with a BRCA1 mutation. Patients will be eligible if they have primary breast cancer (measured on mammogram and ultrasound or MRI) and confirmed histological diagnosis of invasive breast cancer by core biopsy. If axilla lymph nodes will be suspected then fine needle aspiration biopsy will be performed. Patients will be drawn from one of three oncology centers: Szczecin, Bielsko-Biała and Kraków.

Patients will obtain staging investigations and will be monitored. Once entry criteria is met and consent obtained, all patients will obtain baseline staging investigation within 3 weeks of trial registration. Routine investigations will include staging scans: mammography, ultrasound of the breast and axilla (assessment of breast tumor and axilla lymph nodes), assessment of chest/abdomen/pelvis (plain film, Computed Tomography [CT] and/or ultrasound as per local standards) and baseline blood work (Complete Blood Count [CBC], electrolytes, creatinine, Liver Function Tests [LFTs], calcium, albumin).

Once staging investigations are complete, all patients will be treated with cisplatin chemotherapy at a dose of 75mg/m2 every three weeks for a total of four cycles (4 cycles of neoadjuvant chemotherapy). Clinical response will be evaluated every three weeks by the treating physician while on chemotherapy (tumour of the breast and axilla lymph nodes). After four cycles of chemotherapy the patient will then undergo definitive surgery (mastectomy or breast-conserving surgery). Sentinel lymph nodes procedure will be performed. In case of positive lymph nodes standard lymph nodes surgery will be performed. Pathological complete response will defined as no evidence of residual tumor in the breast and the axilla. There may be evidence of ductal carcinoma in situ. The pathology will reviewed by two independent pathologists.

Following surgery patients will receive standard adjuvant chemotherapy at the discretion of the treating physician and if indicated, the patient will also receive radiotherapy and/or hormonal therapy and/or adjuvant trastuzumab at the description of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for enrolment into the trial:

1. Histologically or cytologically proven diagnosis of invasive breast cancer (stage I-III).
2. Documentation of the presence of a germ-line BRCA1 mutation
3. Measurable disease of any size by mammography or ultrasound.
4. Female diagnosed with breast cancer between the ages of 20 to 70.
5. Eastern Cooperative Oncology Group [ECOG] performance status of 0 and 1.
6. Evidence of adequate organ function (liver, bone marrow, kidney)
7. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrolment.
8. Willingness and ability to comply with scheduled visits, treatment plans laboratory tests, and other study procedures.
9. Polish resident.

Exclusion Criteria:

Patients presenting with any of the following will not be included in the trial:

1. Previous chemotherapy for current cancer.
2. Previous or current diagnosis of any other malignancy except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
3. Receiving any medication that may markedly affect renal function.
4. Pregnant or breastfeeding women.
5. Uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-06; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response | Four Months

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Byrski, MD, PhD, Principal Investigator — Pomenarian Medical University
Locations (1):
- Pomenarian Medical University, Szczecin, Poland

REFERENCES:
- [Derived] Byrski T, Huzarski T, Dent R, Marczyk E, Jasiowka M, Gronwald J, Jakubowicz J, Cybulski C, Wisniowski R, Godlewski D, Lubinski J, Narod SA. Pathologic complete response to neoadjuvant cisplatin in BRCA1-positive breast cancer patients. Breast Cancer Res Treat. 2014 Sep;147(2):401-5. doi: 10.1007/s10549-014-3100-x. Epub 2014 Aug 17. PMID 25129345